CLINICAL TRIAL: NCT01287130
Title: A Phase 1 Study of AZD6244 in Combination With Cetuximab in Refractory Solid Tumors
Brief Title: AZD6244 With Cetuximab for Solid Tumors and Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110075; 11-C-0075
Record Dates: First submitted 2011-01-29; First posted 2011-02-01 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-02-05

CONDITIONS: Colonic Neoplasms; Cancer of the Colon; Colon Cancer; Colon Neoplasms; Colonic Cancer
Keywords: Antibodies; Pharmacokinetics; Kinase Inhibitors; Colon Cancer; K-Ras; Colorectal Cancer; Solid Tumor
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Cetuximab; AZD 6244

ARMS (2):
- DL 1 (Experimental): AZD6244 once daily on days 1, 8, 15 and 22. Cetuximab 400 mg/m2 IV loading dose over 120minutes on day 1 and cetuximab 250 mg/m2 IV loading dose over 60 minutes on days 8, 15,22
  Interventions: Drug: Cetuximab; Drug: AZD6244
- DL 2 (Experimental): AZD6244 twice daily on days 1, 8, 15 and 22. Cetuximab 400 mg/m2 IV loading dose over 120minutes on day 1 and cetuximab 250 mg/m2 IV loading dose over 60 minutes on days 8, 15,22
  Interventions: Drug: Cetuximab; Drug: AZD6244

INTERVENTIONS:
Drug: Cetuximab — Day 1 administer cetuximab 400 mg/m2 IV loading dose over 120 minutes. On days 8, 15 and 22 administer cetuximab 250 mg/m2 IV loading dose over 60 minutes
Drug: AZD6244 — Given orally once or twice a day depending on dose level.On days 1, 8, 15 and 22. Repeat every 28 days

SUMMARY:
Background:

- The experimental cancer treatment drug AZD6244 has been shown to block signals that tell cancer cells to grow. Cetuximab, a drug approved to treat cancer of the head, neck, colon, and rectum, also blocks signals that tell cancer cells to grow. Researchers are investigating the highest safe dose of AZD6244 to give with cetuximab, and will also investigate the effectiveness of this drug combination in individuals who have colorectal cancer that involves a particular protein known as the K-RAS protein. Cetuximab is not used to treat colorectal cancer with K-RAS tumors because it has not been shown to be effective, but researchers believe that adding AZD6244 to cetuximab may improve how well cetuximab works, even in people with K-RAS tumors.

Objectives:

* To evaluate the safety and effectiveness of AZD6244 in combination with cetuximab for solid tumors that have not responded to standard treatment.
* To evaluate the safety and effectiveness of AZD6244 in combination with cetuximab for colorectal cancer that involves the K-RAS protein and has not responded to standard treatment.

Eligibility:

* Individuals at least 18 years of age who have been diagnosed with solid tumors that have not responded to standard treatment.
* Individuals at least 18 years of age who have been diagnosed with colorectal cancer that has not responded to standard treatment.

Design:

* This protocol will involve two separate studies: an initial study to establish the highest safe and effective dose of AZD6244 and cetuximab in individuals with solid tumors, and an expansion study of AZD6244 and cetuximab in individuals with colorectal cancer involving the K-RAS protein.
* Participants will be screened with a full medical history and physical examination, blood samples, imaging studies, and other tests as required by the researchers.
* AZD6244 is a capsule to be swallowed once or twice a day, every day, with water on an empty stomach. Cetuximab will be given intravenously once a week, over 2 hours for the first dose and over an hour for every following dose. This combination of daily AZD6244 and weekly cetuximab will be repeated in 28-day cycles of treatment. Participants will keep a diary to record the time of taking AZD6244 each day, as well as any side effects.
* Participants will have frequent blood tests and other exams during the first cycle of treatment, up to five visits to the National Institutes of Health (NIH) and other visits to their local doctor to in the first 28-day cycle.
* During subsequent cycles, participants will have four visits to NIH and four visits to your local doctor for examinations, blood tests, and imaging studies.
* Participants may continue to receive the AZD6244 with cetuximab for up to 6 cycles, until the tumor grows, unacceptable side effects development, or the participant or participant's doctor decides to stop participation. There will be a final study visit that repeats the procedures performed during the screening visit....

DETAILED DESCRIPTION:
Background:

* AZD6244 is an oral highly selective and potent uncompetitive inhibitor of mitogen-activated protein kinase 1/2 (MEK1/2).
* The presence of KRAS mutations predict resistance to EGFR-directed antibody therapy of metastatic colorectal cancer. This appears secondary to KRAS activation of signaling cascades downstream of the EGFR receptor, including the RAF/MEK/ERK pathway.
* Our hypothesis is that EGFR inhibition by cetuximab would be augmented in patients with KRAS mutations if activation of the RAF/MEK/ERK cascade were to be inhibited.

Objectives:

* To determine the dose limiting toxicities and the maximum tolerated dose of AZD6244 in combination with cetuximab in advanced, refractory solid tumors.
* To assess for evidence of anti-tumor activity with this combination, per tumor measurements using RECIST criteria.
* To evaluate the pharmacokinetics of AZD6244 and cetuximab when administered concomitantly.
* To evaluate the safety and tolerability of the combination of AZD6244 and cetuximab in patients with K-RAS mutated metastatic colorectal cancer.
* To assess the inhibition of the RAF/MEK/ERK pathway in peripheral blood mononuclear cells secondary to treatment with AZD6244.
* To evaluate the pharmacokinetics of AZD6244 in combination with cetuximab and the relation to treatment side effects.

Eligibility:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective. In the MTD expansion cohort: Patients must have biopsy proven K-RAS mutant, metastatic colorectal cancer.
* Age greater than or equal to 18
* ECOG performance status less than or equal to 2

Study Design:

* This is a phase 1 dose escalation study of AZD6244 in combination with fixed-dose cetuximab with an expanded cohort in K-RAS mutated metastatic colorectal cancer.
* Patients will be treated with AZD6244 orally twice daily continuously, and cetuximab will be administered at standard doses on days 1, 8, 15 and 22. Dose escalations are outlined per the schema in the parent protocol.
* The dose of AZD6244 will be escalated using a 3-patient cohort design based on first cycle toxicities until dose limiting toxicities (DLT) and maximum tolerated dose (MTD) are defined. Once the MTD/RP2D has been identified, an additional 12 patients with K-RAS mutant colorectal cancer will be enrolled at that dose level, in an effort to more fully characterize pharmacokinetic characteristics of this combination. If at least an 8% response rate is observed in the expanded cohort, the combination will be recommended for future analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:
* In the dose escalation cohorts: Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective. Histology can be based on either the primary tumor or metastases.
* In the MTD expansion cohort: Patients must have biopsy proven K-RAS mutant, metastatic colorectal cancer that has progressed on at least 2 prior standard therapies. K-RAS mutation status must be verified by a CLIA-certified laboratory. (NOTE: colorectal patients enrolled during the dose escalation portion do not need to be K-RAS mutant in order to be eligible).
* Patients must be at least 4 weeks since prior chemotherapy, 6 weeks if the last regimen included nitrosureas or mitomycin C. Prior radiation is allowed as long as the radiation was completed 4 weeks prior to study treatment and no more than 35% of marrow irradiated.
* Age greater than or equal to18 years. Because no dosing or adverse event data are currently available on the use of AZD6244 in combination with cetuximab in patients less than 18 years of age, children are excluded from this study, but will be eligible for future pediatric phase 1 combination trials.
* ECOG performance status less than or equal to 2 (Karnofsky >60%).
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X institutional upper limit of normal (AST and ALT less than or equal to 5.0 X institutional upper limit of normal will be permitted if liver metastases are present)
  * creatinine less than or equal to to to1.5X institution upper limit of normal OR creatinine clearance greater than or equal to 45 mL/min/1.73 m2, as calculated by Cockroft-Gault formula, for patients with creatinine levels above institutional normal. May use a 24 hr. urine collection to determine creatinine clearance.
* Patients may have received prior cetuximab.
* Patients with brain metastases that have been treated and stable for 2 months will be eligible for this study.
* Subjects undergoing anti-coagulation therapy with LMWH and warfarin are eligible. Subjects receiving both warfarin and AZD6244 should have more frequent PT/INR monitoring (see section 10.0)

EXCLUSION CRITERIA:

* Patients who have had chemotherapy, radiotherapy or hormonal therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered (less than or equal to grade 1) from adverse events due to agents administered more than 4 weeks earlier.
* Concurrent treatment with an investigational agent other than the investigational agent(s) used in this study OR treatment within 4 weeks of study entry with any investigational agent(s) or device(s).
* Failure to recover fully (as judged by the investigator) from prior surgical procedures.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244 or other agents used in study.
* Patients taking high doses (more than recommended daily dose) of vitamin E will be excluded. Patients can discontinue use of high dose vitamin E prior to study entry to be considered eligible.
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain AZD6244 capsules.
* Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel are excluded. Subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, prior cardiomyopathy, LVEF less than 50%, unstable angina pectoris, cardiac arrhythmia (i.e. atrial fibrillation), or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because AZD6244 is a small molecule kinase inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD6244, breastfeeding should be discontinued if the mother is treated with AZD6244. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD6244. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients who are serologically positive for Hepatitis B or C, or have a history of liver disease, other forms of hepatitis or cirrhosis are ineligible.
* Use of strong CYP1A2 or 3A4 inducers and/or inhibitors (for example, but not limited to, ketoconazole, rifampacin, atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin (TAO), voriconazole, grapefruit or grapefruit juice, ifabutin, rifapentine, phenytoin, carbamazepine, phenobarbital and St. John's Wort) is not permitted while on study or within 7 days prior to study enrollment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01-07; Primary Completion 2013-08-27 (Actual); Study Completion 2013-08-27 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicities and the maximum tolerated dose of AZD6244 in combination with cetuximab in advanced, refractory solid tumors. | Two year
To assess for evidence of anti-tumor activity with this combination, per tumor measurements | Two year

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of AZD6244 and cetuximab when administered concomitantly | Two years
To evaluate the safety and tolerability of the combination of AZD6244 and cetuximab in patients with K-RAS mutated metastatic colorectal cancer | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Austin G Duffy, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Yeh TC, Marsh V, Bernat BA, Ballard J, Colwell H, Evans RJ, Parry J, Smith D, Brandhuber BJ, Gross S, Marlow A, Hurley B, Lyssikatos J, Lee PA, Winkler JD, Koch K, Wallace E. Biological characterization of ARRY-142886 (AZD6244), a potent, highly selective mitogen-activated protein kinase kinase 1/2 inhibitor. Clin Cancer Res. 2007 Mar 1;13(5):1576-83. doi: 10.1158/1078-0432.CCR-06-1150. PMID 17332304
- [Background] Davies BR, Logie A, McKay JS, Martin P, Steele S, Jenkins R, Cockerill M, Cartlidge S, Smith PD. AZD6244 (ARRY-142886), a potent inhibitor of mitogen-activated protein kinase/extracellular signal-regulated kinase kinase 1/2 kinases: mechanism of action in vivo, pharmacokinetic/pharmacodynamic relationship, and potential for combination in preclinical models. Mol Cancer Ther. 2007 Aug;6(8):2209-19. doi: 10.1158/1535-7163.MCT-07-0231. PMID 17699718
- [Background] Adjei AA, Cohen RB, Franklin W, Morris C, Wilson D, Molina JR, Hanson LJ, Gore L, Chow L, Leong S, Maloney L, Gordon G, Simmons H, Marlow A, Litwiler K, Brown S, Poch G, Kane K, Haney J, Eckhardt SG. Phase I pharmacokinetic and pharmacodynamic study of the oral, small-molecule mitogen-activated protein kinase kinase 1/2 inhibitor AZD6244 (ARRY-142886) in patients with advanced cancers. J Clin Oncol. 2008 May 1;26(13):2139-46. doi: 10.1200/JCO.2007.14.4956. Epub 2008 Apr 7. PMID 18390968
- [Derived] Deming DA, Cavalcante LL, Lubner SJ, Mulkerin DL, LoConte NK, Eickhoff JC, Kolesar JM, Fioravanti S, Greten TF, Compton K, Doyle AG, Wilding G, Duffy A, Liu G. A phase I study of selumetinib (AZD6244/ARRY-142866), a MEK1/2 inhibitor, in combination with cetuximab in refractory solid tumors and KRAS mutant colorectal cancer. Invest New Drugs. 2016 Apr;34(2):168-75. doi: 10.1007/s10637-015-0314-7. Epub 2015 Dec 14. PMID 26666244